CLINICAL TRIAL: NCT06971289
Title: Development and Characterization of Functional Assays for the Analysis of Inflammation Signaling Pathways
Acronym: DEFI
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL25_0250
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Autoinflammatory Disease
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For adult patients:
  3 gel-free heparin tubes and 3 EDTA (EthyleneDiamineTetracetic Acid) tubes during two blood tests as part of routine care
  For Kids :
  depending on Weight
  * Between 12 and 15 kilogram : 1 gel-free heparin tube and 1 EDTA tube during a blood test as part of routine care
  * Between15 and 20 kilogram : 2 gel-free heparin tube and 1 EDTA tube during a blood test as part of routine care
  * Between 20 and 25 kilogram : 2 gel-free heparin tube and 2 EDTA tube during a blood test as part of routine care
  * Between 25 and 30 kilogram: 3 gel-free heparin tube and 2 EDTA tube during a blood test as part of routine care
  * Superior to 30 kg : 3 gel-free heparin tube and 3 EDTA tube during a blood test as part of routine care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood test — blood test as part of routine care

SUMMARY:
Auto-inflammatory diseases are part of a heterogeneous group of illnesses manifested by an inflammatory reaction in its initial phase (innate immunity) that is activated inappropriately: either because the reaction is too strong, or because it is not justified (e.g. in the absence of infection).

Autoinflammatory diseases are often initially described as genetic in origin (i.e. hereditary or familial), and preferentially affect children or young adults. However, the preponderance of auto-inflammation as a cause of symptoms has led to the development of a number of other diseases. In some cases, autoinflammatory diseases may also remain "unclassified".

Generally speaking, autoinflammatory diseases manifest as recurrent attacks of fever, rash and joint pain. Certain signs are more specific to certain diseases, such as urticaria, abdominal pain, mouth ulcers or cervical lymph nodes... It is above all the repetition of the attacks and their unprovoked nature that attract the attention of the patient and the doctor. These attacks are systematically associated with an increase in inflammation markers in the blood.

At present, not all inflammation pathways have been identified. With this study, investigator aim to characterize rare autoinflammatory disease variants and develop relevant cellular models to study inflammation pathways.

ELIGIBILITY:
For adults :

Inclusion Criteria :

* Major patient
* Patient with a rare autoinflammatory disease
* Patient who has given his or her consent to participate in research

Exclusion Criteria :

* Patient under legal protection or safeguard of justice or any other protective measure (guardianship, curatorship)
* Patient with known infection with hepatitis B or C virus or human immunodeficiency virus (HIV)

For Kids :

Inclusion Criteria :

* Minor patients (between 4 and 17 years of age)
* Patient with a rare autoinflammatory disease.
* No additional genetic research will be carried out as part of the project.
* Parents/legal guardians of the child who have given their non-objection to participate in the research.

Exclusion Criteria :

* Patient under legal protection or safeguard of justice or any other protective measure (guardianship, curators)
* Patient with known infection with hepatitis B or C virus or human immunodeficiency virus (HIV)

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with rare autoinflammatory diseases.
  * minor patients, as 70% of rare autoinflammatory diseases are expressed and diagnosed in childhood (Familial Mediterranean Fever (FMF), Periodic Fever-Aphthous Stomatitis-Pharyngitis-Adenopathy Syndrome (PFAPA), Cryopyrin-Associated Periodic Syndrome (CAPS), Mevalonate Kinase Deficiency (MVK)).
  * adult patients, as certain rare autoinflammatory diseases are discovered in adulthood (FMF depending on variant, tumor necrosis factor receptor 1-related relapsing fever syndrome (TRAPS)) or are revealed in adulthood (adult STILL disease, Behçet syndrome, Schnitzler syndrome, VEXAS syndrome (Vacuoles, Enzyme E1, X-linked, Autoinflammatory, Somatic))
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2029-10-15 (Estimated); Study Completion 2029-10-15 (Estimated)

PRIMARY OUTCOMES:
The main judgment criterion will be analysis of the Cytokine/chemokine release assays. | At inclusion Day 0
  Comparison of pro- and anti-inflammatory cytokine concentrations (IL-8, TNF (Tumor Necrosis Factor), chemokine CC ligand 3 and 4 concentrations (CCL3, CCL4) by ELISA in cells supernatants according to the inflammatory pathway involved.